CLINICAL TRIAL: NCT05724277
Title: Comparison of the Effects of Theory of Human Caring Based Short-Term Mindfulness Meditation and Virtual Reality on Patients Scheduled for Laparoscopic Cholecystectomy
Brief Title: The Effect of Mindfulness Meditation and Virtual Reality on Laparoscopic Cholecystectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Seçkin KARAKUŞ, Ataturk University, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SeckinTez
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gall Bladder Disease; Laparoscopic Cholecystectomy
Keywords: recovery; mindfulness; meditation; virtual reality; nursing care
MeSH Terms: conditions — Gallbladder Diseases | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Two different interventions (mindfulness meditation and virtual reality) will be applied to two different experimental groups before surgery. The control group has no intervention.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mindfulness Meditation Group (Experimental): Mindfulness meditation will be applied to the patients in the Mindfulness Meditation Group for 15 minutes in the preoperative period, in both evening and morning.
  Interventions: Behavioral: Mindfulness Meditation
- Virtual Reality Group (Experimental): Virtual reality will be experienced to the patients in the Virtual Reality Group for 15 minutes in the preoperative period, in both evening and morning.
  Interventions: Behavioral: Virtual Reality
- Control Group (No Intervention): The patients in the Control Group will not undergo any intervention in the preoperative period and will receive the routine nursing care of the clinic.

INTERVENTIONS:
Behavioral: Mindfulness Meditation — A 15-minute mindfulness meditation will be conducted by the meditation instructor researcher.
  Arms: Mindfulness Meditation Group
Behavioral: Virtual Reality — A 10-minute virtual reality experience will be provided by using virtual reality glasses.
  Arms: Virtual Reality Group

SUMMARY:
This study aims to compare the effects of the Theory of Human Caring based short-term mindfulness meditation and virtual reality on patients scheduled for laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Anxiety, fear and sleep disorders are frequently encountered conditions in preoperative patient evaluation. Common postoperative problems include pain, sleep disturbances, nausea and vomiting. When these problems are not dealt with effectively, patient comfort and satisfaction are adversely affected, recovery time after surgery and total hospital stay are prolonged, and the time allocated to nursing care increases. Today, it has gained great importance to try to manage these problems with pharmacological and non-pharmacological evidence-based approaches. In particular, nurses need to identify possible problems in both preoperative patient evaluation and postoperative patient follow-up and produce solutions for them. Although it is stated in studies that using easy, effective and safe non-invasive methods such as meditation and virtual reality can reduce the possibility of complications, increase the comfort level of patients, improve the quality of post-surgical recovery, and thus make the surgical process successful, there is no evidence to defend its effectiveness more clearly. more based studies are needed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and over,
* To undergo laparoscopic cholecystectomy operation,
* No orientation problem,
* Volunteering to participate in the study.

Exclusion Criteria:

* Conversion from laparoscopic approach to open cholecystectomy in the operating room,
* Complications that may affect participation in the study,
* Taking the patient to the intensive care unit after surgery,
* Refusal to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
Mindfulness meditation practice provides a positive change in surgical fear in laparoscopic cholecystectomy patients. | the evening before and the morning of the surgery
  In order to evaluate surgical fear, the Surgical Fear Scale will be applied twice, before and after the mindfulness meditation practice, in the preoperative period.
Mindfulness meditation practice provides a positive change in sleep quality in laparoscopic cholecystectomy patients. | in the preoperative period, in the morning of the surgery and in the postoperative period, in the morning after the surgery
  In order to evaluate sleep quality, the Richard Campbell Sleep Questionnaire will be applied in the preoperative period, in the morning of the surgery and in the postoperative period, in the morning after the surgery.
Mindfulness meditation practice provides a positive change in nausea in laparoscopic cholecystectomy patients. | at postoperative 0th, 2nd, 6th, 12th and 24th hours
  In order to evaluate nausea, the Numerical Rating Scale will be applied five times in the postoperative period at the 0th, 2nd, 6th, 12th, and 24th hours after the surgery.
Mindfulness meditation practice provides a positive change in pain in laparoscopic cholecystectomy patients. | at postoperative 0th, 2nd, 6th, 12th and 24th hours
  In order to evaluate the pain, the Numerical Rating Scale will be applied five times in the postoperative period at the 0th, 2nd, 6th, 12th, and 24th hours after the surgery.
Mindfulness meditation practice provides a positive change on the quality of recovery in laparoscopic cholecystectomy patients. | in the preoperative period, evening before surgery and in the postoperative period, morning after surgery
  In order to evaluate the recovery quality, the Quality of Recovery-15T Questionnaire will be applied in the preoperative period and in the postoperative period.
Mindfulness meditation practice provides a positive change on patient satisfaction in laparoscopic cholecystectomy patients. | at 24 hours after surgery
  In order to evaluate patient satisfaction, Watson Caritas Patient Score will be applied once in the postoperative period.
Virtual reality practice provides a positive change in surgical fear in laparoscopic cholecystectomy patients. | the evening before and the morning of the surgery
  In order to evaluate surgical fear, the Surgical Fear Scale will be applied twice, before and after the virtual reality practice, in the preoperative period.
Virtual reality practice provides a positive change in sleep quality in laparoscopic cholecystectomy patients. | in the preoperative period, in the morning of the surgery and in the postoperative period, in the morning after the surgery
  In order to evaluate sleep quality, the Richard Campbell Sleep Questionnaire will be applied in the preoperative period, in the morning of the surgery and in the postoperative period, in the morning after the surgery.
Virtual reality practice provides a positive change in nausea in laparoscopic cholecystectomy patients. | at postoperative 0th, 2nd, 6th, 12th and 24th hours
  In order to evaluate nausea, the Numerical Rating Scale will be applied five times in the postoperative period at the 0th, 2nd, 6th, 12th, and 24th hours after the surgery.
Virtual reality practice provides a positive change in pain in laparoscopic cholecystectomy patients. | at postoperative 0th, 2nd, 6th, 12th and 24th hours
  In order to evaluate pain, the Numerical Rating Scale will be applied five times in the postoperative period at the 0th, 2nd, 6th, 12th, and 24th hours after the surgery.
Virtual reality practice provides a positive change on the quality of recovery in laparoscopic cholecystectomy patients. | in the preoperative period, evening before surgery and in the postoperative period, morning after surgery
  In order to evaluate the recovery quality, the Quality of Recovery-15T Questionnaire will be applied in the preoperative period and in the postoperative period.
Virtual reality practice provides a positive change on patient satisfaction in laparoscopic cholecystectomy patients. | at 24 hours after surgery
  In order to evaluate patient satisfaction, Watson Caritas Patient Score will be applied once in the postoperative period.

SECONDARY OUTCOMES:
Mindfulness meditation and virtual reality applications have positive effects on vital signs. | twice in the preoperative period and five times in the postoperative period
Mindfulness meditation and virtual reality applications have positive effects on blood glucose regulation. | in the preoperative period, morning before surgery and in the postoperative period, morning after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan Binali Yildirim University - Mengücek Gazi Education and Research Hospital, Erzincan, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No